CLINICAL TRIAL: NCT07250594
Title: A Phase II, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multiple-dose Study to Investigate the Safety and Efficacy of 3-month AD17002 Treatment in Adults With Inadequately Controlled Moderate to Severe Eosinophilic Asthma
Brief Title: A Multi-dose Study on the Safety and Efficacy of Self-administered Intranasal AD17002 Treatment for Eosinophilic Asthma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADV-EASP212
Record Dates: First submitted 2025-09-04; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Asthma
Keywords: Eosinophile; Type 1 interferon; Type 2 cytokines; Immunomodulator; eosinophilic asthma; intranasal; self-applicable
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — heat-labile enterotoxin, E coli

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Formulation buffer
  Interventions: Other: Formulation buffer
- Low dose (10 μg) AD17002 (Experimental): containing 10 μg of AD17002
  Interventions: Biological: AD17002
- High dose (20 μg) AD17002 (Experimental): containing 20 μg of AD17002
  Interventions: Biological: AD17002

INTERVENTIONS:
Biological: AD17002 — The IP, AD17002, will be provided in a container, each containing an appropriate number of IP pre-filled, self-administered syringes. Each container will be labeled as required per local requirements
  Arms: High dose (20 μg) AD17002; Low dose (10 μg) AD17002
Other: Formulation buffer — The placebo will be provided in a container, each containing an appropriate volume of formulation buffer, pre-filled syringes for self-administration. Each container will be labeled as required per local requirements
  Arms: Placebo

SUMMARY:
1. Eosinophilic asthma, a type 2 immune disorder, often involves the excessive production of type 2 cytokines.
2. Excessive Type 2 cytokines lead to chronic inflammation, airway hyperresponsiveness, and airflow obstruction.
3. AD17002 is an intranasal self-applicable immunomodulator.
4. AD17002 is safe and tolerable in all studied clinical trials.
5. AD17002 elevates local type-1 interferon levels and promotes epithelial healing.
6. Type-1 interferons have been demonstrated to restore immune balance and reduce eosinophilic infiltration.

AD17002, an innate immune modulator, is likely to be effective as an add-on therapy to control poorly managed moderate to severe eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 on the day of signing the informed consent.
* With a diagnosis of asthma for at least 6 months.
* With pre-BD FEV1 ≥ 50% of the predicted value at the Screening visit (see section 18.6 for calculation of the predicted value for FEV1).
* Having blood eosinophil counts ≥ 150 cells/μL at the Screening visit.
* Participants who meet any of the following asthma criteria at the Screening visit:

  * Moderate asthma-1 (i.e., step 3 in asthma treatment steps in adults and adolescents from 2025 GINA guideline):
  * Moderate asthma-2 (i.e., step 4 in asthma treatment steps in adults and adolescents from 2025 GINA guideline):
  * Severe asthma (i.e., step 5 in asthma treatment steps in adults and adolescents from 2025 GINA guideline, except for biologic therapies):

Exclusion Criteria:

* A current smoker or quit smoking ≤ 0.5 years at Screening visit.
* With serious underlying chronic illness or severe systemic disease, including but not limited to systemic lupus erythematosus, at the investigator's discretion.
* With a current malignancy or previous history of cancer in remission for less than 5 years prior to Screening visit (Subject will not be excluded if he/she had localized carcinoma of the skin that was resected for cure).
* With chronic heart failure in New York Heart Association class III to IV.
* With clinically severe lung disease, including but not limited to cystic fibrosis, chronic bronchitis (chronic obstructive pulmonary disease other than asthma), chronic respiratory infection, lung cancer, current infection, active tuberculosis infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema.
* With arrhythmia, myocardial infarction, or stroke within the last 3 months prior to the Screening visit.
* With a recent respiratory tract infection within 4 weeks prior to the Screening visit.
* Received chronic oxygen therapy within one month prior to the Screening visit.
* With any nasal conditions that could interfere with drug absorption or confound the efficacy or safety assessments.
* Immunosuppressive treatment, including but not limited to methotrexate, troleandomycin, cyclosporine, and azathioprine within 3 months prior to the Screening visit and throughout the study.
* Use of systemic corticosteroids (including regular oral corticosteroids or intramuscular long-acting depot corticosteroids) at daily average doses greater than 7.5 mg prednisone or equivalent for the past 3 months prior to the Screening visit.
* Having or planning to be vaccinated with live (attenuated) vaccine within 1 month prior to the Screening visit and throughout the study.
* Having received immunotherapy including but not limited to monoclonal antibodies, within 3 months prior to the Screening visit and throughout the study.
* Having previously received AD17002.
* Having received other IP or investigational intervention (non-AD17002), including investigational formulations of marketed products, within the past 30 days or 5 half-lives of the medication, whichever is longer, prior to the Screening visit.
* Requiring add-on biologic therapy, such as anti-IgE, anti-IL-5/5R, anti-IL-4Rα, and anti-thymic stromal lymphopoietin treatment.
* Having experienced a life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with high-dose systemic corticosteroids (prednisolone ≥ 40 mg/day or equivalent for ≥ 5 days) within 1 month prior to the Screening visit.
* Having a history of anaphylaxis with cardiorespiratory symptoms, triggered by prior immunotherapy, an unknown cause, or an inhalant allergen.
* Being pregnant or breastfeeding.
* Planning to become pregnant or breastfeed throughout the study.
* A known history of allergy, hypersensitivity, or intolerance to any component of IP, rescue medications, or self-injectable epinephrine.
* Any clinically significant abnormalities in physical examination, vital signs, hematology, biochemistry, or urinalysis that, in the investigator's opinion, may pose a risk to the patient's safety, affect study outcomes, or hinder the patient's ability to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability endpoint | Baseline to week 17
  The incidence and severity of TEAEs and serious TEAEs

SECONDARY OUTCOMES:
Time to the first moderate and severe asthma exacerbations. | Baseline to week 17
  Exacerbation of asthma as defined below:
  Moderate exacerbation of asthma is defined as meeting any one of the following criteria.
  1. Nocturnal awakening(s) for 2 consecutive nights
  2. Daily asthma symptom score Increases ≥ 0.75 from baseline on 2 consecutive days
  3. Increase the use of rescue medication on 2 consecutive days (applicable only when minimum increase: 4 puffs/day)
  4. ≥ 20% decrease in peak expiratory flow (PEF) from baseline on at least 2 consecutive mornings and evenings
  5. Visit to the outpatient department for exacerbation of asthma
  6. ≥ 20% decrease in FEV1 from baseline.
  Severe exacerbation of asthma is defined by any of the following:
  1. Use of systemic corticosteroids, or an increase in the current maintenance dose of oral corticosteroids (OCS), for at least 3 consecutive days.
  2. Emergency department visit, hospitalization, or treatment with systemic corticosteroids due to an acute asthma event.
Proportion of patients experiencing moderate and severe asthma exacerbations | Baseline to week 17
  Exacerbation of asthma as defined below:
  Moderate exacerbation of asthma is defined as meeting any one of the following criteria.
  1. Nocturnal awakening(s) for 2 consecutive nights
  2. Daily asthma symptom score Increases ≥ 0.75 from baseline on 2 consecutive days
  3. Increase the use of rescue medication on 2 consecutive days (applicable only when minimum increase: 4 puffs/day)
  4. ≥ 20% decrease in peak expiratory flow (PEF) from baseline on at least 2 consecutive mornings and evenings
  5. Visit to the outpatient department for exacerbation of asthma
  6. ≥ 20% decrease in FEV1 from baseline.
  Severe exacerbation of asthma is defined by any of the following:
  1. Use of systemic corticosteroids, or an increase in the current maintenance dose of oral corticosteroids (OCS), for at least 3 consecutive days.
  2. Emergency department visit, hospitalization, or treatment with systemic corticosteroids due to an acute asthma event.
Number of moderate and severe asthma exacerbations | Baseline to week 17
  Exacerbation of asthma as defined below:
  Moderate exacerbation of asthma is defined as meeting any one of the following criteria.
  1. Nocturnal awakening(s) for 2 consecutive nights
  2. Daily asthma symptom score Increases ≥ 0.75 from baseline on 2 consecutive days
  3. Increase the use of rescue medication on 2 consecutive days (applicable only when minimum increase: 4 puffs/day)
  4. ≥ 20% decrease in peak expiratory flow (PEF) from baseline on at least 2 consecutive mornings and evenings
  5. Visit to the outpatient department for exacerbation of asthma
  6. ≥ 20% decrease in FEV1 from baseline.
  Severe exacerbation of asthma is defined by any of the following:
  1. Use of systemic corticosteroids, or an increase in the current maintenance dose of oral corticosteroids (OCS), for at least 3 consecutive days.
  2. Emergency department visit, hospitalization, or treatment with systemic corticosteroids due to an acute asthma event.
Time to first asthma worsening alert. | Baseline to week 17
  Asthma worsening alert is defined as any one of the following criteria:
  1. Nocturnal awakening(s) and requiring rescue medication for 2 consecutive nights
  2. Daily symptom score increase of ≥ 0.75 from baseline on 2 consecutive days
  3. Rescue medicine increases from baseline on 2 consecutive days (applicable only when minimum increase: 4 puffs/day)
  4. ≥ 20% decrease in PEF from baseline on at least 2 consecutive mornings and evenings
  5. Outpatient visit for exacerbation of asthma not requiring systemic corticosteroids
  6. ≥ 20% decrease in FEV1 from baseline
Change in pre-bronchodilator (BD) FEV1 | Baseline (Week 1) to Weeks 5, 9, 13, 15, and 17
  FEV1 (Forced Expiratory Volume in 1 Second) is measured using spirometry
Change in FeNO levels | Baseline to week 17
  Fractional Exhaled Nitric Oxide (FeNO) in a clinical trial is measured by an electrochemical FeNO analyzer.
Change in the ratio of weekly average PEF in the morning to predicted PEF from baseline | Baseline to week 17
  The predicted value of PEF equation:
  Men: PEFpred (L/min) = 3.89×Height (cm)-2.95×Age (years)+43.59 Women: PEFpred (L/min) = 4.10×Height (cm)-1.61×Age (years)-173.55 Ratio of PEF = measured weekly average PEF/PEFpred × 100
Change in asthma control | Baseline to week 17
  The ACT is a validated and patient-centric tool (questionnaire) that collects data directly from the patient regarding their symptoms, activity limitations, and medication use. A total of 5 questions. Each question is scored from 1 to 5, and the total is the sum of these scores, with a range of 5 to 25. A score of 19 or less suggests poorly controlled asthma.
Change in blood eosinophil counts | Baseline to week 17
  Measured Blood eosinophil counts (cells/μL)
change in vital signs | Baseline to week 17
  Number of participants with abnormal vital signs.
Change in laboratory values | Baseline to week 17
  Number of participants with abnormal laboratory test results

OTHER OUTCOMES:
Change in percentage of sputum eosinophils | Baseline to week 17
  Measured eosinophil counts in the sputum
Change in serum levels of type 2 cytokines | Baseline to week 17
  Measured by an ELISA-based assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Advagene Biopharma, Taipei, Taiwan, Taiwan